CLINICAL TRIAL: NCT06736730
Title: A Proposal to Establish the Mississippi Violence Injury Prevention (VIP) Program
Brief Title: Mississippi Violence Injury Prevention (VIP) Program
Acronym: MS-VIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: UMMC-IRB-2024-347; 4UH3MD018298-02 (NIH)
Record Dates: First submitted 2024-10-30; First posted 2024-12-17 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Gun Shot Wound
Keywords: Violence prevention; Community-based interventions; Health economics of violence; Clinical trial on violence prevention; Firearm injury prevention; Retaliation and reinjury
MeSH Terms: conditions — Wounds, Gunshot; Reinjuries

STUDY DESIGN:
Intervention Model Description: Jackson, MS will be divided into 9 clusters (with defined geographic boundaries and know population totals) and those clusters will undergo randomization for activation. 3 clusters will be activated each year for three years and those living in the activated clusters will receive the interventions upon activation. Results from participants living in active clusters will be compared to those not in active clusters until at the end of the three years study period all clusters will be activated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Arm (Experimental): Intervention: It includes three key components:
  1. Unrestricted Cash Assistance provided to individuals to support their immediate needs,
  2. Mobile Community Support Services that offer on-site assistance and resources, and
  3. Activation of Operation Good with coordination between hospital and community services to ensure seamless support for individuals affected by violence, promoting recovery and reducing the risk of re-injury or retaliation.
  Interventions: Behavioral: Hospital-Linked Violence Intervention Program; Behavioral: Mobile Community Event Support; Behavioral: Unrestricted Cash Assistance
- In-Active Arm (No Intervention): This group will receive no intervention beyond the standard care provided in the hospital setting. No additional services, cash assistance, or community-based support will be offered. This arm will serve as a comparison group to evaluate the effectiveness of the intervention.

INTERVENTIONS:
Behavioral: Hospital-Linked Violence Intervention Program — Activation of Operation Good, our community partner with a history of direct violence interruption in the streets and longitudinal health and wellness services to firearm injured patient (i.e. linking and aiding those who have suffered from violent injury to mental healthcare, job services, educational services)
  Arms: Active Arm
Behavioral: Mobile Community Event Support — A menu of services provided to the community in an activated cluster where funding will be provided to assist that community in holding events that support overall health and wellness (community clean-up, legal advisory services, pop-up clinic for blood pressure checks).
  Arms: Active Arm
Behavioral: Unrestricted Cash Assistance — A participant in an activated cluster after firearm injury will receive two disbursements of 500$. One at the time of initial hospital evaluation and a second disbursement ~1 month later to offset the financial burden associated with firearm injury on the individual.
  Arms: Active Arm

SUMMARY:
This clinical trial is designed to evaluate the effectiveness of three interventions aimed at preventing violence and supporting those affected by it. Over next three years, the impact of these interventions on key areas will be measured, including the incidence of firearm injuries, the recovery of victims, the occurrence of retaliation and re-injury, and health economics. The interventions are developed based on data collected from a comprehensive needs assessment, community summit, retrospective medical chart reviews, and focus group sessions. The defined interventions are as follows:

Intervention A - Integration of an existing community-based intervention program with Hospital services intervention B - Unrestricted Cash Assistance Intervention C - Mobile Community Support Services

Additionally, the investigators will implement a detailed violence-focused survey for firearm survivors at the time of study enrollment. Follow-up is planned at 3,6 and 12 months. The results of this trial (including analyses of firearm injury rates, recovery outcomes, retaliation/re-injury occurrences, and economic data) will be shared with the affected communities and stakeholders to promote ongoing improvement and support.

DETAILED DESCRIPTION:
To achieve the goals of this trial, the investigators will activate community-focused interventions developed during the first phase of the study to help enroll participants in the study using a stepped wedge cluster design based on their dwelling addresses.

The investigators will formalize the 9 clusters using geographic and demographic data specific to Jackson, Mississippi. Patients presenting in the ER with gunshot injuries will be randomized based on their dwelling address, which will be matched to their corresponding cluster's randomization assignments for the interventions of VIP (Operation Good), Cash Assistance, and Mobile Community Support Services. Any patient with a gunshot injury, regardless of their dwelling address, will be eligible for consent to participate in the longitudinal follow-up of the study. Those not in a currently active clusters at the time of injury will serve as controls for the survey results. Study investigators plan to enroll up to 15 active patients per cluster per year for this follow-up, and community events will be aligned with the same cluster random assignments used for patient interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Firearm injury within the last 24 hours prior to their arrival at the University of Mississippi Medical Center
* Residency/home address within one of the designated clusters.
* Be approached by the research team within 72 hours of arrival.
* Ability to understand the clinical trial, sign the consent form, and commit to follow-ups.
* Ability and willingness to engage in all aspects of the intervention arm (must agree to Operation Good, Survey Participation, and Unrestricted Cash Assistance, these interventions/evaluations cannot be separated)

Exclusion Criteria:

* Self-inflicted gunshot wounds
* Less than 18 years of age
* Patients who are incarcerated or in-custody
* Patients who are unable to understand the clinical trial or sign consent (whether from intoxication, injury, or other cause)
* Patients unable to commit to follow-up or be contacted through routine means

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of death and gunshot injuries | Three years starting upon implementation of the intervention protocol
  The data will be collected from hospital and JPD records. Excluding self-inflicted such as suicide or adjudicated to be accidental/unintentional.

SECONDARY OUTCOMES:
Incidence of PTSD, Score of perceived stress and social cohesion | Three years starting upon implementation of the intervention protocol
  Individual level longitudinal measure and includes "incidence of PTSD, score of perceived stress and social cohesion" collected by individual level surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, PHD, Principal Investigator — Associate Dean For Research And Scholarship
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Formica MK. An Eye on Disparities, Health Equity, and Racism-The Case of Firearm Injuries in Urban Youth in the United States and Globally. Pediatr Clin North Am. 2021 Apr;68(2):389-399. doi: 10.1016/j.pcl.2020.12.009. Epub 2021 Jan 26. PMID 33678293
- [Background] Girling AJ, Hemming K. Statistical efficiency and optimal design for stepped cluster studies under linear mixed effects models. Stat Med. 2016 Jun 15;35(13):2149-66. doi: 10.1002/sim.6850. Epub 2016 Jan 7. PMID 26748662
- [Background] Hooper R, Teerenstra S, de Hoop E, Eldridge S. Sample size calculation for stepped wedge and other longitudinal cluster randomised trials. Stat Med. 2016 Nov 20;35(26):4718-4728. doi: 10.1002/sim.7028. Epub 2016 Jun 28. PMID 27350420
- [Background] Morris MC, Rao U, Garber J. Cortisol responses to psychosocial stress predict depression trajectories: social-evaluative threat and prior depressive episodes as moderators. J Affect Disord. 2012 Dec 20;143(1-3):223-30. doi: 10.1016/j.jad.2012.05.059. Epub 2012 Aug 1. PMID 22858210
- [Background] Zun LS, Downey L, Rosen J. The effectiveness of an ED-based violence prevention program. Am J Emerg Med. 2006 Jan;24(1):8-13. doi: 10.1016/j.ajem.2005.05.009. PMID 16338502
- [Background] Bauer DJ, Preacher KJ, Gil KM. Conceptualizing and testing random indirect effects and moderated mediation in multilevel models: new procedures and recommendations. Psychol Methods. 2006 Jun;11(2):142-63. doi: 10.1037/1082-989X.11.2.142. PMID 16784335
- See also: Mississippi Violence Injury Prevention Program Overview, — https://www.umc.edu/son/MS-VIP